CLINICAL TRIAL: NCT07068035
Title: Investigating the Use of Temporary Abstinence and Expressive Writing for Reducing Problematic Gaming
Brief Title: Effects of Temporary Abstinence and Expressive Writing on Gaming
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Hong Yee Shiun, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NUS-IRB-2023-1037
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Problematic Video Gaming
Keywords: problematic gaming; expressive writing; temporary abstinence; gaming time

STUDY DESIGN:
Intervention Model Description: Participants in the treatment group were instructed to abstain from gaming for a period of 7 days and to engage in expressive writing exercises for 15 minutes every other day for a total of 4 sessions.
  Participants in the control group were instructed to continue their usual gaming routine for a period of 7 days and to engage in control writing exercises for 15 minutes every other day for a total of 4 sessions.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): The treatment group was instructed to abstain from gaming for a period of 7 days and to engage in expressive writing exercises for 15 minutes every other day for a total of 4 sessions
  Interventions: Behavioral: Temporary abstinence and expressive writing
- Control (Other): The control group was instructed to continue their usual gaming routine for a period of 7 days and to engage in control writing exercises for 15 minutes every other day for a total of 4 sessions.
  Interventions: Behavioral: Gaming as per usual and control writing

INTERVENTIONS:
Behavioral: Temporary abstinence and expressive writing — This brief, self-administered intervention combined both temporary gaming abstinence and gaming-focused expressive writing to mitigate gaming problems
  Other Names: temporary abstinence; expressive writing
  Arms: Treatment
Behavioral: Gaming as per usual and control writing — Participants continued with their usual gaming routine and engaged in control writing exercises for 15 minutes every other day for a total of 4 sessions
  Other Names: gaming as per usual; control writing
  Arms: Control

SUMMARY:
The goal of this clinical trial is to investigate if an intervention combining temporary abstinence and expressive writing can mitigate gaming problems in young adult regular gamers. The main questions it aims to answer are:

- Does intervention combining temporary abstinence and expressive writing reduces problematic gaming and gaming time?

Researchers will compare the treatment group to a control group (gaming as per usual and control writing) to examine if the intervention works to mitigate gaming problems.

Participants will:

* Temporarily abstain from video games for a period of 7 days and engage in 4 expressive writing exercises during this intervention period
* Answer three surveys: a baseline survey before the start of the intervention, a post survey after the 7-day intervention, and a follow-up survey 1 month after the post survey.

DETAILED DESCRIPTION:
This clinical trial investigates the effectiveness of a self-administered intervention combining temporary abstinence and expressive writing in addressing problematic gaming behaviours among young adult gamers in Singapore. It aims to evaluate the effectiveness of the intervention in reducing problematic gaming behaviours and improving emotional and health-related outcomes (e.g., psychological distress, physical health status) among young adult gamers by comparing the outcomes among two groups: temporary abstinence with expressive writing group and control group

Participants have to attend an online briefing, complete a baseline survey, take part in a 7-day intervention, complete a post-intervention survey one day later and a 1-month follow-up survey.

1. Online briefing: Participants attended an online briefing session where a member of the research team briefed them on the procedures, emphasised the importance of adhering to the intervention protocol, and addressed any questions that they might have.
2. Baseline survey: Participants were asked to report on their sociodemographics and internet and gaming-related habits, as well as psychosocial characteristics. The baseline survey had to be completed on the same day as the online briefing.
3. Intervention: Participants were randomly assigned to 1 of 2 groups and to take part in the intervention that lasted for 7 consecutive days. In the treatment group, participants were instructed to abstain from gaming for a period of 7 days and to engage in expressive writing exercises for 15 minutes every other day for a total of 4 sessions on Day 1, Day 3, Day 5, and Day 7 of the intervention. Participants typed their writings online using the Qualtrics platform. In the control group, participants were instructed to continue with their usual gaming routine and engaged in control writing exercises for the same number of sessions and duration across the same days.
4. Post-intervention survey: Participants were asked to complete a subset of the baseline survey and a few questions about the intervention (e.g., manipulation checks, compliance).
5. 1-month follow-up survey: Participants were asked to complete a similar set of questionnaires as the baseline survey 1 month after the completion of the post-intervention survey.

ELIGIBILITY:
Inclusion Criteria:

* Singapore citizens/Permanent Residents
* Between 18 and 35 years old
* Play video games regularly (on average at least 7 hours per week)
* Able to read and write English
* Non-professional gamers
* Experience some problems with gaming, use gaming for emotional comfort
* Willing to temporarily take a break from gaming for 7 days

Exclusion Criteria:

* Non-Singapore citizens/Permanent Residents
* Below 18 or above 35 years old
* Do not play video games regularly (less than 7 hours per week)
* Unable to read or write English
* Professional gamers
* Experience no problems with gaming, does not use gaming for emotional comfort
* Unwilling to temporarily take a break from gaming for 7 days

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 321 (Actual)
Dates: Start 2024-08-02 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
problematic gaming | Baseline and 1 month after intervention completion
  Based on the Internet Gaming Disorder Scale-Short-Form. Higher scores indicated greater problematic gaming
gaming hours | Baseline and 1 month after intervention completion
  Participants self-reported the average number of hours spent playing video games per day in a typical week over the past 30 days. This measure quantifies the total time engaged in gaming activity, with higher hours indicating greater gaming engagement.
emotion dysregulation | Baseline, 1 day after intervention completion, and 1 month after intervention completion
  Based on the Difficulties in Emotion Regulation Scale (DERS-18). Higher scores indicated greater emotion dysregulation
maladaptive gaming cognitions | Baseline, 1 day after intervention completion, and 1 month after intervention completion
  Based on the Internet Gaming Cognition Scale. Higher scores indicated greater maladaptive gaming cognitions

SECONDARY OUTCOMES:
psychological distress | Baseline, 1 day after intervention completion, and 1 month after intervention completion
  Based on the Depression, Anxiety and Stress Scale. Higher score indicated greater psychological distress
physical health | Baseline, 1 day after intervention completion, and 1 month after intervention completion
  A single self-report item where participants rated their physical health status at present on a scale from 1 (very poor) to 6 (excellent)
exercise frequency | Baseline, 1 day after intervention completion, and 1 month after intervention completion
  A self-report item where participants reported number of days they engaged in moderate or vigorous physical activity that lasted for more than 10 minutes at a time in a typical week. This item was scored from 1 (never to 1 day per week) to 4 (every day)
sleep quality | Baseline and 1 month after intervention completion
  Based on the Pittsburgh Sleep Quality Index. Higher scores indicated poorer sleep quality

OTHER OUTCOMES:
compensatory behaviours | Baseline, 1 day after intervention completion, and 1 month after intervention completion
  To assess possible compensatory behaviours during intervention period, participants reported the average number of hours that they spent on social media (e.g., Instagram, Facebook, TikTok), watching shows and movies on television and streaming services (e.g., Netflix, Disney+), and browsing gaming-related contents (e.g., game forums) in a typical week

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
The Institutional Review Board's approval is required for the data to be shared. Therefore, IPD that underlie results in a publication are available from the researcher on reasonable request and with the approval of the Institutional Review Board (National University of Singapore)

DOCUMENTS (1):
  • Informed Consent Form (2024-09-23): https://cdn.clinicaltrials.gov/large-docs/35/NCT07068035/ICF_000.pdf